CLINICAL TRIAL: NCT00202696
Title: A Single Center Evaluation of Nalmefene HCl Versus Placebo on Smoking Cessation
Brief Title: Nalmefene Smoking Cessation Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Somaxon Pharmaceuticals (Industry)
Responsible Party: Somaxon Pharmaceuticals, Somaxon Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP-N0408
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2008-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — nalmefene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Nalmefene 40 mg
  Interventions: Drug: nalmefene
- 2 (Experimental): Nalmefene 80 mg
  Interventions: Drug: nalmefene
- 3 (Other): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: nalmefene — Nalmefene HCl film-coated tablets administered orally, twice daily, for total daily dosage of 40 or 80 mg, for 5 weeks (following a 2-week titration period).
  Arms: 1; 2
Other: Placebo — Placebo tablets, administered orally, twice daily for 5 weeks (following a 2-week titration period).
  Arms: 3

SUMMARY:
To determine if nalmefene is safe and effective in smoking cessation.

DETAILED DESCRIPTION:
Single centered, randomized, placebo-controlled,double-blind, outpatient pilot study to evaluate the efficacy, safety and tolerability of 2 doses of nalmefene on smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Smokers in good general health self reporting more than 15 cigarettes per day

Exclusion Criteria:

-

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2005-09; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of 2 doses of nalmefene relative to placebo

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of 2 doses of nalmefene

CONTACTS AND LOCATIONS:
Overall Officials: Philip Jochelson, MD, Study Director — Somaxon Pharmaceuticals CMO
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States